CLINICAL TRIAL: NCT03786458
Title: Development and Evaluation of Web-Based Fertility-Related Decision Support for Young Female Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 201810014RIND
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Infertility, Female; Female Infertility
Keywords: Infertility; young female cancer patients; decision aids; fertility concerns
MeSH Terms: conditions — Infertility, Female; Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cancer and Fertility Decision making (Experimental): Cancer and Fertility Decision aid
  Interventions: Behavioral: web-based decision aid

INTERVENTIONS:
Behavioral: web-based decision aid — The decision aid is then developed further process of evidence synthesis and multidisciplinary external review.

SUMMARY:
This study aims to develop a patient-centered, user-center, interactive web-based decision aid to support the young women with cancer in making an informed fertility-related decision and further evaluate its efficacy.

DETAILED DESCRIPTION:
This study uses mixed-method and involves 2 stages. As following the IPDAS recommendation for developing decision aids, the first sample of 25 young woman survivors with breast, hematology or ovarian cancer, and oncologist, fertility specialists or nurses will be interviewed to assess the fertility-related decision needs from and. The decision aid is then developed further process of evidence synthesis and multidisciplinary external review. After the draft being evaluated for its validity via Think-aloud cognitive interview method, field testing via one-group quasi-experimental design on 90 young women with newly diagnosed breast, hematology or ovarian cancer will be applied to test its outcomes of decision quality, emotional health and fertility concerns.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 to 44
* Have been diagnosed with breast, hematology or ovarian cancer, and will conduct cancer treatment, such as chemotherapy, hormonal or radiation.
* Willing to take questionnaire via computer and tablet.
* Ability to answer the questionnaire with functional emotion and cognition.
* Ability to read newspaper.
* Had been consulted and advised by Doctor on the ability of fertility, but have not decided to give birth to a baby.

Exclusion Criteria:

* Age below 20 or above 45.
* Had been diagnosed with stage 4 cancer.
* Do not require chemotherapy, hormonal or radiation therapy.
* Not able to read newspaper or do not access the internet.

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-08-31 (Estimated); Study Completion 2022-11-27 (Estimated)

PRIMARY OUTCOMES:
Decision conflict,decision regret,fertility knowledge,reproductive concerns after cancer,quality of life | 6 months
  Decisional scale

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Fang Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei City, Taipei, Taiwan